CLINICAL TRIAL: NCT04538118
Title: Relationship of Patient-Specific Functional Scale With Shoulder Functions in Physiotherapy and Rehabilitation Program Applied to Patients With Shoulder Problems
Brief Title: Relationship of Patient-Specific Functional Scale With Shoulder Functions: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 363-37
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Shoulder Impingement; Frozen Shoulder; Humeral Fractures; Rotator Cuff Tears; Disability Physical; Pain, Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome; Bursitis; Humeral Fractures; Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with a shoulder problem: Patients with shoulder problems between 18-65 years of age and being volunteered
  Interventions: Behavioral: Shoulder disability; Device: Shoulder Range of Motion; Behavioral: Pain Intensity

INTERVENTIONS:
Behavioral: Shoulder disability — Shoulder disability was evaluated with Patient-specific functional scale, the disabilities of the shoulder, arm and hand questionnaire, and the upper extremity functional index.
  First assessment was applied when patients came to physical therapy clinic at first.
  Second assessment was repeated after 6 weeks.
Device: Shoulder Range of Motion — Shoulder range of motion was evaluated with universal goniometer. First assessment was applied when patients came to physical therapy clinic at first.
  Second assessment was repeated after 6 weeks.
Behavioral: Pain Intensity — Pain intensity was evaluated with Numeric Pain Rating Scale. First assessment was applied when patients came to physical therapy clinic at first.
  Second assessment was repeated after 6 weeks.

SUMMARY:
The aim of the study is to examine the relationship between the Patient- Specific Functional Scale (PSFS) and shoulder functions in the physiotherapy and rehabilitation program applied to patients with shoulder problems.

ELIGIBILITY:
Inclusion Criteria:

* having a shoulder pathology
* being volunteer
* having shoulder pain at least 3 months
* being literate

Exclusion Criteria:

* having more than one upper extremity pathology
* having an upper extremity pathology involving the neck and trunk
* having a neurological finding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with shoulder problems
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Disability | 6 weeks
  Disability was evaluated with Patient-Specific Functional Scale.Patients nominate 3 to 5 activities that they are unable to do or having difficulty doing because of their injury or problem. These activities are rated on an 11-point scale, where 0 is unable to perform the activity and 10 is able to perform the activity at preinjury level.
Activity Limitation | 6 weeks
  Activity limitation was evaluated with The Disabilities of the Arm, Shoulder and Hand. Scale score ranges from 0 (no disability) to 100 (most severe disability).
Functional Disorder | 6 weeks
  Disability was evaluated with Upper-Extremity Functional Index.Twenty prescribed upper extremity activities are rated by patients according to a 5-point scale, where 0 is extreme difficulty or unable to perform the activity, and 4 is no difficulty. Higher scores mean better outcome scores.

SECONDARY OUTCOMES:
Pain Intensity | 6 weeks
  Pain was evaluated with Numeric Pain Rating Scale. It requires the patient to rate their pain on a defined scale. 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Range of Motion | 6 weeks
  Shoulder range of motion was evaluated with universal goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Hidayet Cuha, MSc, Study Chair — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No